CLINICAL TRIAL: NCT06184451
Title: Effects of TENS During the Performance of a Therapeutic Exercise Protocol in Individuals With Knee Osteoarthritis: Controlled, Randomized, and Blinded Clinical Trial
Brief Title: Effects of TENS During the Performance of a Therapeutic Exercise Protocol in Individuals With Knee Osteoarthritis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Cid André Fidelis de Paula Gomes, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 75610223.5.0000.5511
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise Therapy; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Controlled clinical trial, two arms randomized and blind.
Who Masked: Outcomes Assessor
Masking Description: Two physiotherapists will be responsible for recruiting and assessing inclusion and exclusion criteria. Therefore, a rheumatologist will be responsible for confirming the OA diagnosis of research participants. A researcher will be responsible for the randomization process. Two physiotherapists, blinded to randomization, will be responsible for the assessment procedures. Two other physiotherapists, one for each group, will apply the interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic exercise and Transcutaneous electrical nerve stimulation (Experimental): The therapeutic exercise program includes a warm-up, resistance, neuromuscular, mobility, and balance exercises. Therapeutic exercises will be performed in up to three sets of 8-12 repetitions or 30-60 seconds each, with rest intervals of 90 seconds between sets. Therapeutic exercises will be performed in up to three sets of 8-12 repetitions or 30-60 seconds each, with rest intervals of 90 seconds between sets. TENS will be applied with a portable device during the therapeutic exercise program. The equipment has a two-phase and pulsed symmetric quadratic waveform. 5x5cm adhesive electrodes will be applied to the lateral and medial edges and superior and inferior to the patella, in a crossed manner, surrounding the region.
  Interventions: Other: Therapeutic exercise; Device: Transcutaneous electrical nerve stimulation
- Therapeutic exercise and Placebo Transcutaneous electrical nerve stimulation (Placebo Comparator): Participants in the control group will perform the same therapeutic exercise protocol previously reported in the experimental group, associated with placebo TENS. To do this, the device will only be turned on during the first minute of therapeutic exercises. The same TENS parameters as the experimental group will be applied for this.
  Interventions: Other: Therapeutic exercise; Device: Placebo transcutaneous electrical nerve stimulation

INTERVENTIONS:
Other: Therapeutic exercise — The therapeutic exercise program includes a warm-up, resistance, neuromuscular, mobility, and balance exercises. Therapeutic exercises will be performed in up to three sets of 8-12 repetitions or 30-60 seconds each, with rest intervals of 90 seconds between sets.
Device: Transcutaneous electrical nerve stimulation — TENS will be applied with a portable device, Neurodyn Portable System from Ibramed, while carrying out the entire therapeutic exercise program. The equipment has a two-phase and pulsed symmetric quadratic waveform. 5x5cm adhesive electrodes will be applied to the lateral and medial edges and superior and inferior to the patella, in a crossed manner, surrounding the region.
  The parameters established for the protocol of this study are based on a survey already carried out, with continuous pulse mode, frequency of 150Hz, duration of 150us, and amplitude varying from 1-60mA or more as long as tolerated by the study participant, without causing pain. The application time will be proportional to the time of the exercise session, approximately 60 minutes. The researcher will evaluate the need to adjust the current intensity through the pulse amplitude regularly so that the stimulus does not accommodate.
  Arms: Therapeutic exercise and Transcutaneous electrical nerve stimulation
Device: Placebo transcutaneous electrical nerve stimulation — The equipment has a two-phase and pulsed symmetric quadratic waveform. 5x5cm adhesive electrodes will be applied to the lateral and medial edges and superior and inferior to the patella, in a crossed manner, surrounding the region.
  The parameters established for the protocol of this study are based on a survey already carried out, with continuous pulse mode, frequency of 150Hz, duration of 150us, and amplitude varying from 1-60mA or more as long as tolerated by the study participant, without causing pain. To do this, the device will only be turned on during the first minute of therapeutic exercises. The same TENS parameters as the experimental group will be applied for this.
  Arms: Therapeutic exercise and Placebo Transcutaneous electrical nerve stimulation

SUMMARY:
Research participants diagnosed with knee Osteoarthritis will be randomized through a draw using sealed opaque envelopes indicating two groups: 1. Therapeutic Exercises + Transcutaneous electrical nerve stimulation and 2. Therapeutic Exercises + placebo Transcutaneous electrical nerve stimulation.

Therefore, individuals of both sexes, aged 40 years or over, with a clinical diagnosis of unilateral osteoarthritis of the knee, who present with knee pain for more than three months, morning stiffness for less than 30 minutes, crepitus, bone sensitivity and absence of palpable heat, and diagnosis established radiographically (determined by Kellgren and Lawrence grade 1 to 3 on scale 1 to 4).

Exclusion criteria are bilateral knee Osteoarthritis, hip Osteoarthritis, severe osteoporosis, fibromyalgia, clinical history of tumors or cancer, active inflammatory joint diseases (rheumatoid arthritis, gout), undergoing any lower extremity joint replacement, neurological disorders (Parkinson's disease, stroke, multiple sclerosis, muscular dystrophies, motor neuron disease, Alzheimer's disease), infected wounds or osteomyelitis in the knee region, deep vein thrombosis or thrombophlebitis, sensory changes in the lower limbs, cognitive impairment, and cardiopulmonary disorders that may prevent or limit the execution of exercises, use of a walking assistance device, history of recent trauma to the knee, having undergone any form of treatment involving physiotherapy, intra-articular corticosteroids, anti-inflammatories or chondroprotective within the six months before the start of interventions.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of unilateral osteoarthritis of the knee
* presenting knee pain for more than three months
* morning stiffness for less than 30 minutes
* crepitus, bone tenderness, and absence of palpable heat.

Exclusion Criteria:

* Bilateral knee osteoarthritis, hip osteoarthritis
* severe osteoporosis
* fibromyalgia
* medical history of tumors or cancer
* active inflammatory joint diseases (rheumatoid arthritis, gout),
* undergoing any lower extremity joint replacement
* neurological diseases (Parkinson's disease, Accident Cerebral Vascular, Multiple Sclerosis, muscular dystrophies, motor neuron disease, Alzheimer's disease)
* infected wounds or osteomyelitis in the knee region
* deep vein thrombosis or thrombophlebitis
* sensory changes in the lower limbs
* cognitive and cardiopulmonary impairment that may prevent or limit performing the exercises
* using a walking assistance device
* having a history of recent trauma to the knee,
* having undergone any form of treatment involving physiotherapy
* intra-articular corticosteroids, anti-inflammatories, or chondroprotective in the six months before the start of the interventions.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Functional disability | Change from Baseline, after 5 weeks of intervention and 4 weeks after the end of the intervention.
  Knee Injury and Osteoarthritis Outcome Score (KOOS). It aims to evaluate the domains of pain, symptoms, activities of daily living, function related to recreation and sports, and quality of life related to the knee. Totaling 42 items, each item must be answered using a Likert scale that ranges from 0 (best score) to 4 (worst score), and the score for each subscale ranges from 0 (worst score) to 100 (best score).

SECONDARY OUTCOMES:
Numerical Pain Scale | Change from Baseline, after 5 weeks of intervention and 4 weeks after the end of the intervention.
  The Numerical rating pain scale, a simple, easily administered scale evaluates the perceived intensity of pain, using an 11-point scale from 0, representing 'no pain', to 10, which is the 'worst possible pain'.
Functional self-perception | Change from Baseline, after 5 weeks of intervention and 4 weeks after the end of the intervention.
  Pain self-efficacy questionnaire, structured into 10 items where each item is evaluated by selecting a number on a 7-point numerical scale (scores from 0 to 6), where 0 means "not at all confident" and 6 means "completely confident". The items cover different functions, from work, social activities, domestic tasks and coping with pain without medication. A total score is calculated from the sum of the scores for each of the 10 items, producing a total score that ranges from 0 to 60. Higher scores reflect stronger self-efficacy beliefs.
Lower limb functionality | Change from Baseline, after 5 weeks of intervention and 4 weeks after the end of the intervention.
  30 second sit and stand test. From a sitting position with feet flat on the floor and shoulder-width apart, arms crossed across the chest, the individual assessed must stand, with hips and knees fully extended. Then, he must sit down, with his lower part completely touching the seat, repeating these movements continuously for 30 seconds. The chair must be placed against the wall. The total number of complete cycles will be counted (standing up and sitting down represents one cycle).
Self-perceived functionality | Change from Baseline, after 5 weeks of intervention and 4 weeks after the end of the intervention.
  Patient Specific Functional Scale. An easy-to-apply self-report instrument, validated for measuring disability related to specific tasks identified by the individual. The scale is made up of 11 (eleven) numbers, graduated from 0 (zero) to 10 (ten), where 0 (zero) represents inability to perform the activity and ten (ten) the ability to perform the activity at the level prior to the current condition.
Maximum voluntary isometric contraction | Change from Baseline, after 5 weeks of intervention and 4 weeks after the end of the intervention.
  manual dynamometer portable (Lafayette Manual Muscle System, Modelo 01165, Lafayette Instrument Company, Lafayette, IN). Four 5-second readings will be taken during maximal voluntary isometric contraction (MVIC) with a 30-second rest period between contractions. The first CIVM will familiarize the volunteer with carrying out the task. A new set of readings will be taken if a volunteer can perform three contractions with at least 10% variability. Strong and constant verbal stimuli will be used throughout the test. Always with the research participants' hands positioned crossed on the chest. Thus, bilateral assessments of the muscles, quadriceps, and gluteus medius will be carried out. The order of CIVM readings will be randomized to avoid collection bias. The research participant will remain in lateral decubitus with a pillow positioned between the legs, with the limb to be tested superiorly in a neutral position.
Global Perception of Change scale | Change from Baseline, after 5 weeks of intervention and 4 weeks after the end of the intervention.
  The perception of the global effect of the treatment by the research participant will be evaluated by the Global Perception of Change scale. The Global Perception of Change scale is a direct scale on the patient's self-perception when the intervention is performed. This scale consists of 11 points, ranging from -5 (worsening compared to the start of treatment), 0 (neutral) and +5 (improvement compared to the start of treatment), using the Portuguese version.
Functionality | Change from Baseline, after 5 weeks of intervention and 4 weeks after the end of the intervention.
  The World Health Organization Disability Assessment Schedule 2.0 short version (12 items) is a generic self-report assessment instrument developed by the World Health Organization (WHO) to assess functionality and disability during the last 30 days.For each item, a Likert-type scale will be used to define the severity of the limitation, with a score of 0 (Zero) denoting "no limitation" and 4 (four) denoting "extreme limitation or inability to function." The total score is the sum of all 12 items, where a score of 48 points represents the worst possible restriction.

CONTACTS AND LOCATIONS:
Overall Officials: Cid Gomes, PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- Nove de Julho University, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Make data available remotely in digital cloud storage.